CLINICAL TRIAL: NCT04812171
Title: Healing of Apical Periodontitis After Nonsurgical Endodontic Treatment- the Effect of Diabetes Mellitus and Tobacco Smoking
Brief Title: Healing of Apical periodontitis-the Effect of Diabetes Mellitus and Tobacco Smoking
Status: Completed | Type: Observational
Sponsor: Romana Peršić Bukmir (Other)
Collaborators: University of Rijeka (Other)
Responsible Party: Sponsor-Investigator, Romana Peršić Bukmir, Ph.D., University Hospital Rijeka
Organization: University Hospital Rijeka (Other)
Other Study IDs: Uniri-biomed-18-53 1183
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Periapical Periodontitis
Keywords: Diabetes mellitus; Periapical periodontitis; Smoking
MeSH Terms: conditions — Periapical Periodontitis; Diabetes Mellitus; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- smoker participants: Current cigarette smokers older than 18 years, without previously reported systemic disease, not taking medications influencing imunological system or bone metabolism.
  Received adequate endodontic treatment of at least one tooth and attending follow-up at six months and one year following root-canal treatment.
  Interventions: Procedure: non-surgical endodontic treatment
- non-smoker participants: Healthy non-smokers paired with smoker group according to age and gender. Received adequate endodontic treatment of at least one tooth and attending follow-up at six months and one year following root-canal treatment.
  Interventions: Procedure: non-surgical endodontic treatment
- diabetic participants: Participants reporting diabetes melitus type II, having gycated hemoglobin test, not taking medications influencing imunological system or bone metabolism, non-smokers Received adequate endodontic treatment of at least one tooth and attending follow-up at six months and one year following root-canal treatment.
  Interventions: Procedure: non-surgical endodontic treatment
- non-diabetic participants: Healthy non-smokers paired with diabetic group according to age and gender. Received adequate endodontic treatment of at least one tooth and attending follow-up at six months and one year following root-canal treatment.
  Interventions: Procedure: non-surgical endodontic treatment

INTERVENTIONS:
Procedure: non-surgical endodontic treatment — standard non-surgical endodontic treatment performed by endodontic specialist

SUMMARY:
Apical periodontitis is an inflammatory process located around the apex of the root. It is mainly caused by a microbial infection of the pulp space. Diabetes mellitus and tobacco smoking are modulating factors that may influence the healing of apical periodontitis. Present studies have disclosed an association between smoking and apical periodontitis and diabetes mellitus and apical periodontitis. The aim of this study is to compare the healing of periapical bone in smokers and non-smokers and patients with diabetes mellitus type 2 and healthy participants. The hypothesis of this study is that smokers and patients diagnosed with diabetes mellitus will experience slower healing with a lower success rate in comparison to control groups. Apical periodontitis will be diagnosed through means of clinical examination and radiological analysis. Healing of apical periodontitis will be determined using periapical radiographs utilizing periapical index. This prospective study will contribute to the development of clinical guidelines concerning smokers and patients with diabetes mellitus type 2.

DETAILED DESCRIPTION:
Apical periodontitis is an inflammatory process located around the apex of the root. It is mainly caused by a microbial infection of the pulp space. Diabetes mellitus and tobacco smoking are modulating factors that may influence the healing of apical periodontitis. Present studies have disclosed an association between smoking and apical periodontitis and diabetes mellitus and apical periodontitis. The aim of this study is to compare the healing of periapical bone in smokers and non-smokers and patients with diabetes mellitus type 2 and healthy participants. The hypothesis of this study is that smokers and patients diagnosed with diabetes mellitus will experience slower healing with a lower success rate in comparison to control groups. Apical periodontitis will be diagnosed through means of clinical examination and radiological analysis. Healing of apical periodontitis will be determined using periapical radiographs utilizing periapical index (PAI). One observer will be calibrated by evaluation of periapical status in 100 reference radiographs according to periapical index scoring system .

In each participant only one tooth will be included in the study. This will be first tooth submitted to endodontic treatment according to diagnostic priority. The survey will include only teeth with adequate endodontic treatment according to following criteria: post-operative periapical radiograph demonstrating adequate length and homogeneity of root canal filling (no visible voids, one millimeter shorter than radiologic apex) , and clinically and radiologically adequate permanent crown restoration. Participants will attend clinical and radiological follow-up in six months and one year following root-canal treatment to assess healing rate. In diabetic participants glycemic control will be determined according to the level of glycated hemoglobin, which is routine procedure in these patients. In smokers, intensity and duration of smoking habit will be recorded. This prospective study will contribute to the development of clinical guidelines concerning smokers and patients with diabetes mellitus type 2.

ELIGIBILITY:
Inclusion Criteria

1. Influence of smoking habit on apical periodontitis healing after non-surgical endodontic treatment

   * Smoker group- everyday cigarette smoking habit, older than 18 years
   * Control group-healthy non-smoker patients, older than 18 years, paired with smoker group according to age and sex
2. Influence of diabetes mellitus on apical periodontitis healing after non-surgical endodontic treatment

   * Diabetic group-patients having type 2 diabetes mellitus, older than 18 years, non-smokers
   * Control group-healthy patients, non-smokers, older than 18 years, paired with diabetic group according to age and sex

Exclusion Criteria:

1. Influence of smoking habit on apical periodontitis healing after non-surgical endodontic treatment

   * Smoker group-systemic disease, pregnancy, taking medications that interfere with bone metabolism and immunologic response, former and occasional smokers
   * Control group-former, occasional and present smokers,systemic disease, pregnancy, taking medications that interfere with bone metabolism and immunologic response
2. Influence of diabetes mellitus on apical periodontitis healing after non-surgical endodontic treatment Diabetic group-pregnancy, taking medications that interfere with bone metabolism and immunologic response, smokers Control group-patients having diabetes mellitus, pregnancy, taking medications that interfere with bone metabolism and immunologic response, smokers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort of patients attending Dental Clinic of the Rijeka Clinical Hospital Centre requiring root canal treatment of at least one tooth with radiological diagnosis of apical periodontitis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Influence of smoking habit on apical periodontitis healing after non-surgical endodontic treatment | one year
  Comparison of apical periodontitis healing in smoker and non-smoker participants
Influence of diabetes mellitus on apical periodontitis healing after non-surgical endodontic treatment | one year
  Comparison of apical periodontitis healing in diabetic and non-diabetic participants

SECONDARY OUTCOMES:
Association of smoking intensity and duration with apical periodontitis healing | one year
  Calculation of association of smoking intensity and duration with apical periodontitis healing rate
Association of glycated hemoglobin level (HbA1C) with apical periodontitis healing | one year
  Calculation of association of glycated hemoglobin level (HbA1C) with apical periodontitis healing rate

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Pezelj-Ribarić, PhD,DMD, Study Director — Faculty of Dental Medicine, University of Rijeka, Croatia
Locations (1):
- University of Rijeka Faculty of Dental Medicine, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: Undecided